CLINICAL TRIAL: NCT07351851
Title: Effects of PEMM in Chronic Low Back Pain Women With Urinary Incontinence A Randomised Controlled Trial
Brief Title: Effects of PEMM in Chronic Low Back Pain Women With Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Manisha Pramod Shenoy, Clinician: Physiotherapy Specialist, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRC-01-24-698
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-09

CONDITIONS: Chronic Low-back Pain (cLBP); Urinary Incontinence (UI); Pelvic External Myofascial Mobilisation; Myofascial Techniques; Pelvic Pain
Keywords: chronic low back pain; urinary incontinence; myofascial mobilisation; PEMM; female pelvic pain
MeSH Terms: conditions — Urinary Incontinence; Pelvic Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: The study will involve recruiting women having UI and CLBP. Patients meeting the inclusion criteria will be randomly allocated in experimental and control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Reassessment will be done on the 8th week where the outcome measures of pain, SF36, ODI, ICIQ-UI-SF will be recorded. an independent assessor will be assigned for the recording. the assessor will not have access to the inital recording of outcome measure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEMM (Experimental): PEMM therapy with theragun and strengthening for 6 weeks duration.
  Interventions: Other: PEMM with Theragun
- Control (Active Comparator): TENS and hot pack for 15 min, symptomatic pain treatment with strengthening for 6 weeks duration.
  Interventions: Other: Active Comparator: Control

INTERVENTIONS:
Other: PEMM with Theragun — PEMM will be given with theragun at specific assessed points and strengthening exercises will be given
  Other Names: Pelvic External Myofascial Mobilisation
  Arms: PEMM
Other: Active Comparator: Control — Pain modulation will be given with TENS and hot pack, and strengthening exercises will be given
  Other Names: TENS and strengthening
  Arms: Control

SUMMARY:
Urinary incontinence (UI), Chronic low back pain (CLBP) in women are prevalent and often coexist. Multiple conditions when coexist, it leads to reduced Quality of life in turn causing physical and mental impairment. Musculoskeletal structures and fascial restrictions is one of the attribute to the coexistence of urinary incontinence and chronic back pain in women. External myofascial mobilization (EMM) with core exercises have been proven beneficial for conditions in males that is caused by musculoskeletal and fascial structures. However there are limited research which proves the effect of EMM in conditions involving musculoskeletal and fascial structures . Therefore, the aim of the study is to find the effect of MFTs in reducing the disability in women with CLBP and UI PRIMARY OBJECTIVE To evaluate the effectiveness of PEMM treatment in reducing disability, pain and improving mental health in women with CLBP and UI Study design : Simple randomization Sampling method: Simple Random sampling Random numbers will be generated in Excel, then random numbers will be presented in a concealed envelope for the participants to choose Sample Size : 130 (Experimental 65, Control 65) Sample size was determined using expected effect size i.e., mean change in the primary outcome variable disability index reported in the recent research study . With effect size (change in the disability index score) 3.5 and standard deviation of the change in the outcome 6.45, statistical power 80% and level of significance 5%, the required sample size would be n=55 participants in each group. However, to accounts for multiple secondary outcome measures, possible dropouts and non-response it would be good to increase an additional 20% in calculated sample size i.e., a total of 130 participants (65 participants in each group) will be included in this study.

The following sample size equation was used to determine adequate sample size:n = [2 (Z?/2 + Z?)2 * ?2] / (m1-m2)2 Where Z? and Z? are the values standard normal variate e.g., at 5% level of significance Z?/2 = 1.96, and with 80% power the value of Z?= 0.84; ? is the polled Standard deviation and m1 and m2 are the mean outcome values s in group 1 and group 2 respectively.

Blinding:

Single blinding: patient will be blinded to the group allocation. The assessor is blinded to the treatment

Material and tools :

Theragun - Theragun Elite, 20 V, Myofascial tools - foam roll, foam ball, Questionnaires - SF 3642,43,44, Oswestry Low back pain questionnaire (ODI)45 and The International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI-SF)46 PROCEDURE In the course of the study the total number of patients referred to physiotherapy department with LBP will be interviewed to identify patients with or without UI having LBP. The data obtained from this will be recoded as prevalence in results. The documents of the patients having LBP with UI will be reviewed to check who fulfills the inclusion criteria. All who meets the inclusion criteria will be approached face to face with the aim of the study. Informed consent form will be given to patients who are volunteering to participate in the study. The data of the participants who do not wish to participate in the study will also be recorded.

The participants who have consented to participate in the study will be then assessed. Since the participants has UI she will be directed to a Urologist for an assessment. After urologist assessment, patients will be randomly allocated to experimental and control groups. Random allocation will be administered by the random numbers generated and will be presented in a concealed envelope for the participants to choose. 1st week, the demographic data and Outcome measure of pain, SF36, ODI, ICIQ-UI-SF will be recorded (1st time) on the day of assessment. The outcome measures will be printed on paper and will be given to the patients to fill up with a pen, all questionnaires are self reported outcome measures. Treatment will commence a week after, where experimental group will undergo PEMM therapy with strengthening for 6 weeks duration and the control group will have conventional symptomatic pain treatment with strengthening (2nd to 7th week). Treatment will be given for 6 weeks (1 sessions in a week). The treatment day may vary any day between 4th and 7th day post one session. After 6 sessions of treatment, patient will be advised HEP (Home exercise program) to continue at home. Reassessment will be done on the 8th week where the outcome measures of pain, SF36, ODI, ICIQ-UI-SF will be recorded. Participants will be educated and advised regarding HEP. Exercises will be taught to the patient by explanation, demonstration, teach-back method, and printed sheet of exercise. Compliance to HEP will be recorded before final Outcome measure

ELIGIBILITY:
Inclusion Criteria:

* Age group of 18 - 65 years
* Has child/children <5 parity
* CLBP patients with UI referred for physiotherapy for CLBP
* Patient with low back pain for more than 3 months
* NRS more than 5/10
* Patient with complain of urinary incontinence since past 3 months or more

Exclusion Criteria:

* Chronic Low Back Pain with red flags
* Not able to read and write in English /Arabic
* Pregnant ladies and post partum 1 year
* UTI, Pelvic floor Surgery
* Any systemic condition of renal and cardiac
* Patient with active carcinoma or any inflammatory disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females only
Enrollment: 200 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
VAS Pain | Week 1 and week 8
  Visual analogue scale
Oswestry disability index | Week 1 and week 8
urinary incontinence scale | Week 1 and week 8
  ICIQ-UI-SF - International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form

SECONDARY OUTCOMES:
mental and physical quality of life | Week 1 and week 8
  SF 36

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Baladīyat ad Dawḩah, Qatar

IPD SHARING:
Plan to Share IPD: Undecided
I will be happy to share it if the organisation i am working under allows me.

REFERENCES:
- [Result] Ajimsha MS, Ismail LA, Al-Mudahka N, Majzoub A. Effectiveness of external myofascial mobilisation in the management of male chronic pelvic pain of muscle spastic type: A retrospective study. Arab J Urol. 2021 Jul 26;19(3):394-400. doi: 10.1080/2090598X.2021.1954414. eCollection 2021. PMID 34552791
- [Result] Park SH, Kang CB. Effect of Kegel exercises on the management of female stress urinary incontinence: a systematic review of randomized controlled trials. Advances in Nursing. 2014
- [Result] .Lin, A., Abbas, H., Sultan, M., & Tzeng, T. (2022). A critical review of interventional treatments for myofascial pelvic pain. Journal of the International Society of Physical and Rehabilitation Medicine,
- [Result] Tozzi P, Bongiorno D, Vitturini C. Fascial release effects on patients with non-specific cervical or lumbar pain. J Bodyw Mov Ther. 2011 Oct;15(4):405-16. doi: 10.1016/j.jbmt.2010.11.003. Epub 2011 Jan 8. PMID 21943614
- [Result] Lin, A., Abbas, H., Sultan, M., & Tzeng, T. (2022). A critical review of interventional treatments for myofascial pelvic pain. Journal of the International Society of Physical and Rehabilitation Medicine
- [Result] Pool-Goudzwaard A, van Dijke GH, van Gurp M, Mulder P, Snijders C, Stoeckart R. Contribution of pelvic floor muscles to stiffness of the pelvic ring. Clin Biomech (Bristol). 2004 Jul;19(6):564-71. doi: 10.1016/j.clinbiomech.2004.02.008. PMID 15234479
- [Result] Hodges PW, Sapsford R, Pengel LH. Postural and respiratory functions of the pelvic floor muscles. Neurourol Urodyn. 2007;26(3):362-71. doi: 10.1002/nau.20232. PMID 17304528
- [Result] Sapsford RR, Hodges PW. Contraction of the pelvic floor muscles during abdominal maneuvers. Arch Phys Med Rehabil. 2001 Aug;82(8):1081-8. doi: 10.1053/apmr.2001.24297. PMID 11494188
- [Result] Radebold A, Cholewicki J, Panjabi MM, Patel TC. Muscle response pattern to sudden trunk loading in healthy individuals and in patients with chronic low back pain. Spine (Phila Pa 1976). 2000 Apr 15;25(8):947-54. doi: 10.1097/00007632-200004150-00009. PMID 10767807
- [Result] Hodges PW, Richardson CA. Inefficient muscular stabilization of the lumbar spine associated with low back pain. A motor control evaluation of transversus abdominis. Spine (Phila Pa 1976). 1996 Nov 15;21(22):2640-50. doi: 10.1097/00007632-199611150-00014. PMID 8961451
- [Result] Barr KP, Griggs M, Cadby T. Lumbar stabilization: a review of core concepts and current literature, part 2. Am J Phys Med Rehabil. 2007 Jan;86(1):72-80. doi: 10.1097/01.phm.0000250566.44629.a0. PMID 17304690
- [Result] Mogren IM, Pohjanen AI. Low back pain and pelvic pain during pregnancy: prevalence and risk factors. Spine (Phila Pa 1976). 2005 Apr 15;30(8):983-91. doi: 10.1097/01.brs.0000158957.42198.8e. PMID 15834344
- [Result] Welk B, Baverstock R. Is there a link between back pain and urinary symptoms? Neurourol Urodyn. 2020 Feb;39(2):523-532. doi: 10.1002/nau.24269. Epub 2020 Jan 3. PMID 31899561
- [Result] Cassidy T, Fortin A, Kaczmer S, Shumaker JTL, Szeto J, Madill SJ. Relationship Between Back Pain and Urinary Incontinence in the Canadian Population. Phys Ther. 2017 Apr 1;97(4):449-454. doi: 10.1093/ptj/pzx020. PMID 28339852
- [Result] Mutaguchi M, Murayama R, Takeishi Y, Kawajiri M, Yoshida A, Nakamura Y, Yoshizawa T, Yoshida M. Relationship between low back pain and stress urinary incontinence at 3 months postpartum. Drug Discov Ther. 2022;16(1):23-29. doi: 10.5582/ddt.2022.01015. PMID 35264471
- [Result] Bertuit J, Bakker E, Rejano-Campo M. Relationship between urinary incontinence and back or pelvic girdle pain: a systematic review with meta-analysis. Int Urogynecol J. 2021 May;32(5):1073-1086. doi: 10.1007/s00192-020-04670-1. Epub 2021 Feb 23. PMID 33620534
- [Result] Dal Farra F, Aquino A, Tarantino AG, Origo D. Effectiveness of Myofascial Manual Therapies in Chronic Pelvic Pain Syndrome: A Systematic Review and Meta-Analysis. Int Urogynecol J. 2022 Nov;33(11):2963-2976. doi: 10.1007/s00192-022-05173-x. Epub 2022 Apr 7. PMID 35389057
- [Result] Stuge B. Pelvic girdle pain: examination, treatment, and the development and implementation of the European guidelines. Journal of the Association of Chartered Physiotherapists in Womens Health. 2012
- [Result] Borenstein DG. Chronic low back pain. Rheum Dis Clin North Am. 1996 Aug;22(3):439-56. doi: 10.1016/s0889-857x(05)70281-7. PMID 8844907
- [Result] Meucci RD, Fassa AG, Faria NM. Prevalence of chronic low back pain: systematic review. Rev Saude Publica. 2015;49:1. doi: 10.1590/S0034-8910.2015049005874. Epub 2015 Oct 20. PMID 26487293
- [Result] Alzahrani H, Mackey M, Stamatakis E, Zadro JR, Shirley D. The association between physical activity and low back pain: a systematic review and meta-analysis of observational studies. Sci Rep. 2019 Jun 3;9(1):8244. doi: 10.1038/s41598-019-44664-8. PMID 31160632
- [Result] Endresen EH. Pelvic pain and low back pain in pregnant women--an epidemiological study. Scand J Rheumatol. 1995;24(3):135-41. doi: 10.3109/03009749509099301. PMID 7777823
- [Result] Ghafouri A, Alnaimi AR, Alhothi HM, Alroubi I, Alrayashi M, Molhim NA, Shokeir AA. Urinary incontinence in Qatar: A study of the prevalence, risk factors and impact on quality of life. Arab J Urol. 2014 Dec;12(4):269-74. doi: 10.1016/j.aju.2014.08.002. Epub 2014 Sep 10. PMID 26019961
- [Result] Lukacz ES, Santiago-Lastra Y, Albo ME, Brubaker L. Urinary Incontinence in Women: A Review. JAMA. 2017 Oct 24;318(16):1592-1604. doi: 10.1001/jama.2017.12137. PMID 29067433
- [Result] Stothers L, Friedman B. Risk factors for the development of stress urinary incontinence in women. Curr Urol Rep. 2011 Oct;12(5):363-9. doi: 10.1007/s11934-011-0215-z. PMID 21938471
- [Result] Reynolds WS, Dmochowski RR, Penson DF. Epidemiology of stress urinary incontinence in women. Curr Urol Rep. 2011 Oct;12(5):370-6. doi: 10.1007/s11934-011-0206-0. PMID 21720817
- [Result] Aoki Y, Brown HW, Brubaker L, Cornu JN, Daly JO, Cartwright R. Urinary incontinence in women. Nat Rev Dis Primers. 2017 Nov 16;3:17097. doi: 10.1038/nrdp.2017.97. PMID 29143807
- [Result] Alghadir AH, Tse C, Iqbal A, Al-Khater M, Al-Rasheed G. The Prevalence and Association of Stress Urinary Incontinence, Core Muscle Endurance, and Low Back Pain among Married Women in Saudi Arabia: A Case-Control Study. Biomed Res Int. 2021 Jul 15;2021:5533241. doi: 10.1155/2021/5533241. eCollection 2021. PMID 34337021